CLINICAL TRIAL: NCT02515240
Title: Immune Response to Pneumococcal Vaccination in HIV Infected Individuals
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIV PPV23; 5R01AI081558 (NIH)
Record Dates: First submitted 2015-07-07; First posted 2015-08-04 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Pneumococcal Infection
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- healthy controls (Active Comparator): healthy individuals, HIV negative, 19-50 yrs if age, immunized with one shot of PPV23 vaccine.
  Interventions: Biological: PPV23
- newly diagnosed HIV >200 (Active Comparator): Newly diagnosed HIV positive patients with CD4 count >200, immunized with one shot of PPV23 vaccine.
  Interventions: Biological: PPV23
- newly diagnosed HIV <200 (Active Comparator): Newly diagnosed HIVpositive patients with CD4 count <200, immediately immunized with one shot of PPV23 vaccine.
  Interventions: Biological: PPV23
- newly diagnosed HIV <200 delayed (Active Comparator): Newly diagnosed HIV positive patients with CD4 count <200 delayed immunization with one shot of PPV23 vaccine, treated for 6-12 months with Highly Active Anti-Retroviral Therapy (HAART) first.
  Interventions: Biological: PPV23
- HAART experienced HIV>200 (Active Comparator): HIV positive, on HAART treatment for 5 years, nadir CD4 count <200, but at present CD4 count is >200, immunized with one shot of PPV23 vaccine.
  Interventions: Biological: PPV23
- HAART experienced HIV<200 (Active Comparator): HIVpositive, on HAART treatment for 5 years, nadir CD4 count <200, and at present CD4 count is <200, immunized with one shot of PPV23 vaccine.
  Interventions: Biological: PPV23

INTERVENTIONS:
Biological: PPV23 — 23 valent pneumococcal polysaccharide vaccine in Healthy adults.
  Other Names: 23 valent pneumococcal polysaccharide vaccine

SUMMARY:
The purpose of the study. To characterize the immune response to the pneumococcal vaccine in HIV positive individuals and to dissect the most appropriate timing and frequency of vaccination.

DETAILED DESCRIPTION:
All potential study candidates will be asked to fill out a questionnaire concerning their medical history and medications. This survey will determine eligibility. If eligible, as part of the experimental protocol the HIV positive participants will agree to be randomized to immediate vs. delayed pneumococcal immunization and 3 blood draws around the time of immunization. The HIV negative control population will agree to immunization with pneumococcal polysaccharide vaccine (PPV), not standard of care for this population, and 3 blood draws around the time of immunization. The investigators will study the effect of pneumococcal vaccination in HIV positive adults. At the present time it is recommended that all HIV positive individuals receive the pneumococcal vaccine at the time of diagnosis with those with cluster of differentiation (CD4) count <200 to be vaccinated either immediately or alternatively, treated with highly active antiretroviral therapy (HAART) for 6 months followed by PPV. All patients are recommended to be re-vaccinated at 5 years. This is the standard of care. It is however unclear how the HIV positive patients respond to PPV. In the 1st part of the study, Part I, newly diagnosed HIV positive individuals will be recruited. As standard of care, these individuals will receive the pneumococcal vaccine regardless of their participation in this study. Those that agree to participate in the study will be grouped according to their CD4 count: >500, 200-500 or <200. Those with a CD4 count <200 will be randomly assigned to receive the vaccine immediately or to receive HAART for 6 months prior to vaccination, this is in accordance with the present recommendations, either immediate vaccination or giving HAART for 6 months prior to vaccination is considered acceptable.. Thus ALL HIV positive individuals will receive the vaccine as presently recommended. The HIV positive volunteers agree to (experimental part of the protocol):

1. Be randomized to either immediate vaccination vs. 6 months after start of HAART if the CD4 count is <200
2. Donate blood specimens at 3 different times: day 0, day of vaccination: 2 mL, at day 7, 40 mL and at day 28-42 a one time sample of 2 mL.
3. Have their blood samples subjected to antibody analysis (concentration and functional activity) and antibody gene usage analysis There will be 4 HIV positive groups in this part of the study: CD4>500, CD4 200-500, CD4 < 200 immediate vaccination and CD4 <200, delayed vaccination.

There will be 19 individuals per group. The HIV negative controls in Part I of the study (n=19) who agree to participate will also be vaccinated with the pneumococcal vaccine. This is NOT a vaccine recommended for healthy adults but is NOT contra-indicated.

Thus as part of the experimental procedure for these individuals they will:

1. Receive the FDA approved pneumococcal vaccine
2. Blood samples will be obtained at day 0: 2 mL, day 7 40 mL and day 28-42, one time sample of 2 mL.
3. Blood samples will be analyzed for antibody concentration, functional activity and gene family usage.

In summary, we will study a total of 5 groups in Part I:

Group 1: HIV positive CD4>500 Group 2: HIV positive CD4 200-500 Group 3: HIV positive CD4 < 200 immediate vaccination Group 4: HIV positive CD4<200 delayed (6 months) vaccination Group 5: HIV negative In part II of the study the investigators will evaluate the effect of a second pneumococcal vaccination, which is presently recommended, in HIV positive individuals, to be received 5 years after the first vaccination. Again, only those HIV positive individuals who are due for their second pneumovax will be asked to participate. They will be grouped according to their CD4 counts as CD4 >500 or CD4 200-500. Thus ALL HIV positive individuals will receive the vaccine as recommended.

The HIV positive volunteers solely agree to;

1. Donate blood specimens at 3 different occasions: day 0, day of vaccination: 2 mL, at day 7, 40 mL and at day 28-42 a one time sample of 2 mL.
2. Have their blood samples subjected to antibody analysis (concentration and functional activity) and antibody gene usage analysis There will be 2 HIV positive groups: CD4>500 and CD4 count 200-500. There will be 19 individuals per group.

The HIV negative controls in Part II of the study who agree to participate will be recruited from the population of individuals previously vaccinated with pneumovax. They will also be vaccinated for the second time with the pneumococcal vaccine, 5 years after the first vaccination. This is NOT a vaccine recommended for healthy adults but is NOT contra-indicated. Thus as part of the experimental procedure for these individuals they will:

1. Receive the FDA approved pneumococcal vaccine
2. Blood samples will be obtained at day 0: 2 mL, day 7 40 mL and day 28-42 one time sample of 2 mL.
3. Blood samples will be analyzed for antibody concentration, functional activity and gene family usage.

In summary, we will study 3 groups in Part II of the study Group 6: HIV positive CD4>500, 2nd PPV Group 7: HIV positive CD4 200-500, 2nd PPV Group 8: HIV negative, 2nd PPV.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative:
* never immunized with PPV23
* HIV positive:
* need for PPV23 per standard of care

Exclusion Criteria:

* steroid use
* other immunosuppressive agents;
* pregnancy
* incapable of completing consent form

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2010-07; Primary Completion 2014-06 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Antibody activity and response by opsonophagocytic assay (OPT) and ELISA (ug/ml) | Day 0 and day 30 of vaccination

SECONDARY OUTCOMES:
Polysaccharide-specific B cell phenotype: percentage naive or memory B cell distribution flow cytometry | Day 0 and Day7 of vaccination
Flow cytometry : percentage cells expressing tumor necrosis factor receptors on surface | Day 0 and Day7 of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Julie MA Westerink, MD, Principal Investigator — University of Toledo-HSC
Locations (1):
- The University of Toledo-Health Science Campus, Toledo, Ohio, United States

REFERENCES:
- [Result] Ballet JJ, Sulcebe G, Couderc LJ, Danon F, Rabian C, Lathrop M, Clauvel JP, Seligmann M. Impaired anti-pneumococcal antibody response in patients with AIDS-related persistent generalized lymphadenopathy. Clin Exp Immunol. 1987 Jun;68(3):479-87. PMID 3652522
- [Result] Janoff EN, Douglas JM Jr, Gabriel M, Blaser MJ, Davidson AJ, Cohn DL, Judson FN. Class-specific antibody response to pneumococcal capsular polysaccharides in men infected with human immunodeficiency virus type 1. J Infect Dis. 1988 Nov;158(5):983-90. doi: 10.1093/infdis/158.5.983. PMID 3183430
- [Result] Klein RS, Selwyn PA, Maude D, Pollard C, Freeman K, Schiffman G. Response to pneumococcal vaccine among asymptomatic heterosexual partners of persons with AIDS and intravenous drug users infected with human immunodeficiency virus. J Infect Dis. 1989 Nov;160(5):826-31. doi: 10.1093/infdis/160.5.826. PMID 2572650
- [Result] Kroon FP, van Dissel JT, Ravensbergen E, Nibbering PH, van Furth R. Enhanced antibody response to pneumococcal polysaccharide vaccine after prior immunization with conjugate pneumococcal vaccine in HIV-infected adults. Vaccine. 2000 Nov 22;19(7-8):886-94. doi: 10.1016/s0264-410x(00)00232-2. PMID 11115712
- [Result] Loeliger AE, Rijkers GT, Aerts P, Been-Tiktak A, Hoepelman AI, van Dijk H, Borleffs JC. Deficient antipneumococcal polysaccharide responses in HIV-seropositive patients. FEMS Immunol Med Microbiol. 1995 Sep;12(1):33-41. doi: 10.1111/j.1574-695X.1995.tb00171.x. PMID 8580899
- [Result] Ochs HD, Junker AK, Collier AC, Virant FS, Handsfield HH, Wedgwood RJ. Abnormal antibody responses in patients with persistent generalized lymphadenopathy. J Clin Immunol. 1988 Jan;8(1):57-63. doi: 10.1007/BF00915157. PMID 2966810
- [Result] Opravil M, Fierz W, Matter L, Blaser J, Luthy R. Poor antibody response after tetanus and pneumococcal vaccination in immunocompromised, HIV-infected patients. Clin Exp Immunol. 1991 May;84(2):185-9. doi: 10.1111/j.1365-2249.1991.tb08146.x. PMID 2025948
- [Result] Ragni MV, Ruben FL, Winkelstein A, Spero JA, Bontempo FA, Lewis JH. Antibody responses to immunization of patients with hemophilia with and without evidence of human immunodeficiency virus (human T-lymphotropic virus type III) infection. J Lab Clin Med. 1987 May;109(5):545-9. PMID 3572201
- [Result] Rodriguez-Barradas MC, Musher DM, Lahart C, Lacke C, Groover J, Watson D, Baughn R, Cate T, Crofoot G. Antibody to capsular polysaccharides of Streptococcus pneumoniae after vaccination of human immunodeficiency virus-infected subjects with 23-valent pneumococcal vaccine. J Infect Dis. 1992 Mar;165(3):553-6. doi: 10.1093/infdis/165.3.553. PMID 1347058
- [Result] Unsworth DJ, Rowen D, Carne C, Sonnex C, Baglin T, Brown DL. Defective IgG2 response to Pneumovax in HIV seropositive patients. Genitourin Med. 1993 Oct;69(5):373-6. doi: 10.1136/sti.69.5.373. PMID 8244356
- [Result] Berberian L, Goodglick L, Kipps TJ, Braun J. Immunoglobulin VH3 gene products: natural ligands for HIV gp120. Science. 1993 Sep 17;261(5128):1588-91. doi: 10.1126/science.7690497.
- [Result] Berberian L, Shukla J, Jefferis R, Braun J. Effects of HIV infection on VH3 (D12 idiotope) B cells in vivo. J Acquir Immune Defic Syndr (1988). 1994 Jul;7(7):641-6. PMID 8207642
- [Result] Karray S, Zouali M. Identification of the B cell superantigen-binding site of HIV-1 gp120. Proc Natl Acad Sci U S A. 1997 Feb 18;94(4):1356-60. doi: 10.1073/pnas.94.4.1356. PMID 9037057
- [Result] Townsley-Fuchs J, Neshat MS, Margolin DH, Braun J, Goodglick L. HIV-1 gp120: a novel viral B cell superantigen. Int Rev Immunol. 1997;14(4):325-38. doi: 10.3109/08830189709116523. PMID 9186784
- [Result] Muller S, Kohler H. B cell superantigens in HIV-1 infection. Int Rev Immunol. 1997;14(4):339-49. doi: 10.3109/08830189709116524. PMID 9186785
- [Result] Chang Q, Abadi J, Alpert P, Pirofski L. A pneumococcal capsular polysaccharide vaccine induces a repertoire shift with increased VH3 expression in peripheral B cells from human immunodeficiency virus (HIV)-uninfected but not HIV-infected persons. J Infect Dis. 2000 Apr;181(4):1313-21. doi: 10.1086/315405. Epub 2000 Apr 13. PMID 10762563
- [Derived] Iyer AS, Khaskhely NM, Leggat DJ, Ohtola JA, Saul-McBeth JL, Khuder SA, Westerink MA. Inflammatory Markers and Immune Response to Pneumococcal Vaccination in HIV-Positive and -Negative Adults. PLoS One. 2016 Mar 1;11(3):e0150261. doi: 10.1371/journal.pone.0150261. eCollection 2016. PMID 26930208